CLINICAL TRIAL: NCT04642352
Title: Office-Based Superior Laryngeal Nerve (SLN) Block for Treatment of Neurogenic Cough
Brief Title: Office-Based Superior Laryngeal Nerve Block for Treatment of Neurogenic Cough
Status: Recruiting | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Blake Simpson, Principal Investigator, University of Alabama at Birmingham
Other Study IDs: IRB-300005783
Record Dates: First submitted 2020-11-19; First posted 2020-11-24 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Cough
Keywords: chronic cough
MeSH Terms: conditions — Cough; Chronic Cough | interventions — Bupivacaine; Triamcinolone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- SLN intervention group: Participants will undergo a superior laryngeal nerve (SLN) block
  Interventions: Drug: superior laryngeal nerve block

INTERVENTIONS:
Drug: superior laryngeal nerve block — A unilateral injection of 2 cc of a 1:1 mixture of 0.25% bupivacaine and Kenalog-40 via a 27 gauge needle to the thyrohyoid space (front of neck, just above larynx/voice box) via a 27 gauge needle to the thyrohyoid space (front of neck, just above larynx/voice box) on the side which exhibited most discomfort/tenderness/cough on palpation. If neither side was uncomfortable, the right side will be used.
  Other Names: 0.25% bupivacaine; Kenalog-40

SUMMARY:
The purpose of this study is to evaluate if office-based injection of a local anesthetic/steroid combination at the area of one superior laryngeal nerve can decrease cough frequency and alleviate symptoms of chronic cough in patients with neurogenic cough.

DETAILED DESCRIPTION:
Neurogenic cough is a chronic cough without a clear cause. It is thought to be related to irritation of a nerve that goes to the larynx (voice box). This can happen after a viral upper respiratory infection. Current treatment uses therapy or medications taken by mouth. Those medications can be sedating and not well tolerated. An alternative approach would be to perform an injection "nerve block", which is commonly done for other nerve disorders such as around the spine. This may help people with neurogenic cough also. We studied this recently in a small group of patients and found that patients had improvement in their cough symptoms (Simpson 2018). It would be helpful to study this in a larger group of patients using more methods of evaluating cough symptom severity.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Ability of patients to speak and understand English
* Ability for patients to consent for themselves
* Cough for 8 weeks or greater, with suspected sensory neuropathic etiology of the cough. Inclusion based on history of preceding upper respiratory infection or other symptoms suggestive of irritable larynx such as cough in response to temperature changes, odors, scents/perfumes, tickle, irritation in the throat/paralaryngeal region, or talking.
* Persistent cough despite treatment of ALL the major contributors of cough (items listed below would be done as part of a standard clinical workup for chronic cough and are not done specific to this study):

  * Reflux disease treatment with one of the following: failure of two months of PPIs OR negative pH study
  * Asthma: lack of response to at least one month of steroid inhaler/bronchodilator OR normal PFTs/negative methacholine challenge + negative CXR/CT
  * Upper airway cough syndrome/Allergic disease: lack of response to at least one month of antihistamines/decongestants/nasal steroids OR negative allergy testing (skin or serum) OR lack of response to at least one year of immunotherapy/allergy shots

Exclusion Criteria:

* Age less than 18 years
* Patients unable or unwilling to provide informed consent
* Known etiology to cough other than sensory neuropathy (e.g., reflux disease, asthma, allergic rhinitis, chronic obstructive pulmonary disease)
* Addition of new neuromodulators at the time of the injection. Patients who were already being treated with neuromodulators for their cough (e.g., gabapentin, amitriptyline) will not be excluded provided their dose remains constant.
* Nissen fundoplication within the last year
* Smoking history within last 5 years
* Allergy to bupivacaine or Kenalog-40

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to UAB Department of Otolaryngology for the evaluation and treatment of chronic cough who would be undergoing superior laryngeal nerve block as part of their standard clinical care.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-01-03 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Change in score on the Leicester Cough Questionnaire | Baseline to 3 months
  The Leicester Cough Questionnaire consists of 19 questions designed to assess the impact of cough on various aspects of a participant's quality of life. Scores are chosen from a Likert scale from 1 to 7, with 1 representing "all of the time" and 7 representing "none of the time." Scores would decrease if symptoms improved.

CONTACTS AND LOCATIONS:
Overall Officials: Blake Simpson, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No